CLINICAL TRIAL: NCT00864630
Title: Objective Detection, Evaluation and Countermeasures for In-flight Depression
Brief Title: Neuroimaging for Depression
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study upon which this project depended for subjects and the intervention was terminated prematurely due to lack of funds.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Emory University (Other)
Responsible Party: Gary Strangman, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NSBRI-NBFP01301
Record Dates: First submitted 2009-03-17; First posted 2009-03-19 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2011-05

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wait list (No Intervention)
- Computer-based problem solving therapy (Experimental)
  Interventions: Behavioral: Computer-based problem solving therapy

INTERVENTIONS:
Behavioral: Computer-based problem solving therapy — Computer program developed by Dr. James Cartriene at Beth Israel Deaconess Hospital, Boston, MA.
  Arms: Computer-based problem solving therapy

SUMMARY:
The investigators seek to determine whether brain imaging techniques can be used to help detect depression, assess its severity, and/or monitor or predict responses to treatment. Subjects with minor or major depression will be randomly assigned to a wait-list control group or to treatment with a new computer-based cognitive behavior therapy developed by Dr. James Cartriene. Brain imaging will be performed before and during treatment using both magnetic resonance imaging (MRI) and near-infrared spectroscopy (NIRS). The investigators hypothesize that brain activity, particularly in the lateral frontal areas of the brain, will provide biomarkers for depression, depression severity, and treatment response.

DETAILED DESCRIPTION:
Depression can significantly disrupt one's ability to function effectively and efficiently, and the associated performance deficits can seriously jeopardize space mission success. The incidence of serious depression in Earth based analogues of the spaceflight environment has been reported as up to 13% per person per year. Extrapolating from existing reports of depressive episodes during short-duration spaceflight, depression is thus a probable condition in one or more members of a five to seven person crew during a long duration spaceflight (e.g., a 30 month mission to Mars). Mission success can be jeopardized by depression either directly, from the potentially life threatening consequences of lapses in performance, or indirectly, by adding to the workload and stress of other crewmembers. The likelihood and potentially serious consequences of depression during spaceflight explains why the risk of human performance failure due to mood alterations such as depression, anxiety, or other psychiatric and cognitive problems is a Priority 1 risk for all mission types (International Space Station, Moon, Mars). Certain countermeasures are already in place: medications and psychological consultations with ground-crews. However, current in-flight methods to decide whether a countermeasure should be used rely heavily on subjective self-reports. The biological basis of mood disorders suggests neural biomarkers may provide a more objective method for assessing depression. Aim 1 of this proposal, therefore, seeks to identify neural biomarkers sensitive to, and specific for, depression. These measures will be used in evaluating and validating a flight-capable, noninvasive neuroimaging technology (near-infrared spectroscopy and imaging, or NIRS imaging) for its ability to detect biomarkers of depression and its severity. As an initial step towards developing novel select-out criteria, Aim 2 will then evaluate which neural biomarkers appear most promising in detecting an endophenotype that identifies individuals at heightened risk for treatment resistance. Finally, when depression is objectively identified, an appropriate countermeasure needs to be selected. Aim 3 will focus on the ability of brain imaging to help predict the efficacy of Dr. Cartriene's computer based problem solving therapy.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV criteria for minor or major depression
* Written informed consent
* Age 30-60 years (age of individuals currently in the astronaut corps)

Exclusion Criteria:

* Suicidal or homicidal ideation
* Women who are pregnant, breastfeeding, or women of childbearing potential who are not using a medically accepted means of contraception
* Known history of serious or unstable medical illness
* History of seizure disorder, brain injury, any history of known neurological disease
* Clinical or lab evidence of untreated hypothyroidism
* History or DSM-IV diagnosis of organic mental disorder, schizophrenia, schizoaffective disorder, delusional disorder, psychotic disorders not otherwise specified, bipolar disorder, patients with mood congruent or mood incongruent psychotic features, patients with substance use disorders (excluding alcohol and nicotine) active within the last 12 months
* Current use of other psychotropic drugs, including current use of benzodiazepines, hypnotics, anticonvulsants
* Patients who have failed to respond during the course of their current major depressive episode to at least two antidepressant trials
* Currently undergoing depression-focused psychotherapy
* Patients who have taken an investigational psychotropic drug within the past year
* Patient cannot safely enter the MRI scanning environment
* Latex allergy

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-10 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Functional magnetic resonance imaging | Pre-therapy and 4 weeks after therapy initiation

SECONDARY OUTCOMES:
Functional near infrared neuroimaging | Pre-therapy and 2 and 4 weeks after therapy initiation
MRI-based brain perfusion | Pre-therapy and 4 weeks after therapy initiation
MRI-based brain morphology | Pre-therapy and 4 weeks after therapy initiation
MRI-based diffusion imaging | Pre-therapy and 4 weeks after therapy initiation

CONTACTS AND LOCATIONS:
Overall Officials: Gary E Strangman, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States